CLINICAL TRIAL: NCT04904627
Title: Constructive Variations of Classic Orthopedic Braces for Spinal Deformity During Growth: Efficacy Analysis of a Retrospective Cohort
Brief Title: Constructive Variations of Classic Orthopedic Braces for Spinal Deformity During Growth
Status: Recruiting | Type: Observational
Sponsor: Istituto Scientifico Italiano Colonna Vertebrale (Other)
Responsible Party: Sponsor
Other Study IDs: COB-ISICO
Record Dates: First submitted 2021-05-12; First posted 2021-05-27 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Polyehtylene vs Poliìycarbonate: super rigid vs rigid material
- Free pelvis vs classic pelvis: fixed pelvis versus free pelvis, allowing adjustment in the sagittal plane.

SUMMARY:
The construction methods of the same brace vary on an experiential basis according to who builds them, the prescriber, the characteristics of the patients and also the innovations introduced to ensure greater comfort for the patient. The closure of the brace or the way in which the two shells are fixed varies at the discretion of the orthopedic technician. Plastic materials have also changed. In addition, the use of the classic cast for the production of the negative model was gradually replaced by cad-cam technology. In some cases, modular constructions were introduced with respect to the customized one. All this has changed the classic corsets over time, even without changing their name / type, and according to the hypothesis that their effectiveness remained at least the same, if not even improved.

There are no publications that have shown variations in efficacy that can be correlated with some of these stylistic variations.

The purpose of this study is to retrospectively investigate whether the various innovations and stylistic variations over time have had an effect on the clinical, functional and radiographic outcomes in growing subjects suffering from spinal deformity treated with corsets at a specialized center.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic adolescent scoliosis and/or dorsal hyperkyphosis,
* age under 16 years at the start of observation,
* brace prescription for more than 18 hours/day,
* availability of radiographs of the entire spine while standing and in brace radiographs at 1 month or out of brace at 5 ± 2 months at the end growth after 48 hours without brace and at 1 year.
* availability of compliance data
* Risser between 0 and 4 at first assessment

Exclusion Criteria:

* All secondary causes of scoliosis
* history of spinal fusion surgery
* lack of one of the radiographic examinations required by the protocol

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Growing subjects suffering from spinal deformity (adolescent idiopathic scoliosis and / or hyperkyphosis) undergoing brace treatment.
Sampling Method: Non-Probability Sample
Enrollment: 470 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changes in radiographic measurements | pre-treatment, in brace after a month from the start of wearing and without brace after 5 ± 2 months, after an average period of 4 years +/-2 , after 48 hours without brace and 1 year later.
  variation of Cobb degrees of the main curve in the frontal plane over time
Changes in radiographic measurements | pre-treatment, in brace after a month from the start of wearing and without brace after 5 ± 2 months, after an average period of 4 years +/-2 , after 48 hours without brace and 1 year later.
  variation of Cobb degrees of all curves in the frontal and sagittal plane over time.

SECONDARY OUTCOMES:
HRQOL | pre-treatment, after a month from the start of brace wearing, after 5 ± 2 months, after an average period of 4 years +/-2 , and 1 year later
  measures of quality of life. The Italian Spine Youth Quality of Life questionnaire (ISYQOL) measures the health-related quality of life of adolescents with spinal deformities. ISYQOL consists of 20 items, each scored 0, 1 or 2. In accordance with the Rasch analysis technique, used to develop the questionnaire, the ordinal ISYQOL total score is converted to an interval measure (i.e., ISYQOL measure), which is expressed on a 0%-100% scale (with 100% indicating high quality of life).
HRQOL | pre-treatment, after a month from the start of brace wearing, after 5 ± 2 months, after an average period of 4 years +/-2 , and 1 year later
  measures of quality of life. The Scoliosis Research Society-22 (SRS-22) is a questionnaire developped to measure health-related quality of life in patients with idiopathic scoliosis. It has 22 questions divided into five domains: function/activity, pain, self-image/appearance, mental health and satisfaction with management. Each domain contains five questions, except the satisfaction with management domain, which contains two questions. Each item can be scored from 1 (worst possible) to 5 (best possible). The function/activity, pain, self-image and mental health domains have a total score ranging from 5 to 25. The satisfaction with management domain has a total score ranging from 2 to 10. The maximum total score is 110 and the results are expressed as a mean
Treatment outcome | after an average period of 4 years +/-2
  variation of the main curve of at least 5 Cobb degrees, end treatment results: main curve </=30 Cobb degrees, main curve </=45 Cobb degrees, and main curve >50 Cobb degrees
Treatment compliance | after a month from the start of brace wearing, after 5 ± 2 months, and after an average period of 4 years +/-2
  Treatment compliance measures: percentage of brace wearing declared and measured by heat sensors
Deformity clinical measures | pre-treatment, after a month from the start of brace wearing, after 5 ± 2 months,after an average period of 4 years +/-2 , and 1 year later
  score on the evaluation of the aesthetic profile of the trunk (TRACE)
Deformity clinical measures | pre-treatment, after a month from the start of brace wearing, after 5 ± 2 months,after an average period of 4 years +/-2 , and 1 year later
  measurement of the hump on the Adams test in degrees
Deformity clinical measures | pre-treatment, after a month from the start of brace wearing, after 5 ± 2 months,after an average period of 4 years +/-2 , and 1 year later
  measurement of the hump on the Adams test in millimeters

CONTACTS AND LOCATIONS:
Locations (1):
- ISICO, Milan, Mi, Italy